CLINICAL TRIAL: NCT05724654
Title: Longer-term Effects of Peanut Consumption on Brain Function in Older Men and Women
Brief Title: Effects of Peanut Consumption on Brain Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: The Peanut Institute Foundation (TPIF) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: METC 22-046
Record Dates: First submitted 2023-01-11; First posted 2023-02-13 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Brain Vascular Function; Cerebral Blood Flow; Brain Insulin Sensitivity; Cognitive Performance

STUDY DESIGN:
Intervention Model Description: Study participants will receive in random order daily 60 g of skin roasted peanuts (peanut intervention) or no peanuts for a total of 16 weeks (control intervention), separated by a wash-out period of at least 8 weeks.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Skin roasted peanuts
  Interventions: Dietary Supplement: Skin roasted peanuts
- Control (No Intervention): No skin roasted peanuts

INTERVENTIONS:
Dietary Supplement: Skin roasted peanuts — Study volunteers will receive daily 60 g of skin roasted peanuts for 16 weeks.
  Arms: Experimental

SUMMARY:
Impaired brain vascular function precedes the development of reduced cognitive performance, while brain insulin-resistance is also associated with cognitive decline. Peanut consumption has already been shown to beneficially affect cognitive performance. However, underlying mechanisms have not yet been established, while well-controlled trials on longer-term effects of peanuts on cognitive performance are highly needed. The hypothesis is that longer-term peanut consumption has beneficial effects on (regional) cerebral blood flow responses (primary outcome), which may relate to an improved cognitive performance (secondary outcome) in older men and women. Important objectives are to investigate in older adults the effect of 16-week peanut consumption on (i) brain vascular function in cognitive-control brain areas, and (ii) brain insulin-sensitivity. We will also focus on changes in cognitive performance as assessed with a neuropsychological test battery (secondary objective). Cerebral blood flow responses before (brain vascular function) and after the administration of intranasal insulin (brain insulin-sensitivity) will be quantified by the non-invasive gold standard magnetic resonance imaging (MRI)-perfusion method Arterial Spin Labeling (ASL).

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged between 60-75 years
* BMI between 20-35 kg/m2
* Fasting plasma glucose < 7.0 mmol/L
* Fasting serum total cholesterol < 8.0 mmol/L
* Fasting serum triacylglycerol < 4.5 mmol/L
* Systolic blood pressure < 160 mmHg and diastolic blood pressure < 100 mmHg
* Stable body weight (weight gain or loss < 3 kg in the past three months)
* Willingness to give up being a blood donor from 8 weeks before the start of the study, during the study and for 4 weeks after completion of the study
* No difficult venipuncture as evidenced during the screening visit

Exclusion Criteria:

* Allergy or intolerance to peanuts
* Left-handedness
* Current smoker, or smoking cessation < 12 months
* Diabetic patients
* Familial hypercholesterolemia
* Abuse of drugs
* More than 3 alcoholic consumptions per day
* Use of products or dietary supplements known to interfere with the main outcomes as judged by the principal investigators
* Use medication to treat blood pressure, lipid, or glucose metabolism
* Use of an investigational product within another biomedical intervention trial within the previous 1-month
* Severe medical conditions that might interfere with the study, such as epilepsy, asthma, kidney failure or renal insufficiency, chronic obstructive pulmonary disease, inflammatory bowel diseases, auto inflammatory diseases, and rheumatoid arthritis
* Active cardiovascular disease like congestive heart failure or cardiovascular event, such as an acute myocardial infarction or cerebrovascular accident
* Contra-indications for MRI imaging (e.g., pacemaker, surgical clips/material in body, metal splinter in eye, claustrophobia)

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Brain Vascular Function | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  Cerebral blood flow as quantified non-invasively by the MRI perfusion method Arterial Spin Labeling (ASL)
Brain Insulin Sensitivity | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  Change in cerebral blood flow, as quantified non-invasively by the MRI perfusion method Arterial Spin Labeling (ASL), before and after application of intranasal insulin (160 IU)

SECONDARY OUTCOMES:
Cognitive Performance | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  Cambridge Neuropsychological Test Automated Battery (CANTAB)

OTHER OUTCOMES:
Brain Perfusion | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  Transcranial Doppler (TCD) ultrasound will be used to assess the velocity of blood flow through the middle cerebral artery (MCA)
Retinal Microvasculature | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  Retinal images made by fundus camera
Systolic Blood Pressure | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  Office blood pressure
Diastolic Blood Pressure | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  Office blood pressure
Heart Rate | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  Heart rate measured during office blood pressure measurement
Circulating Lipids and Lipoproteins | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  High-Density Lipoprotein (HDL) cholesterol, Low-Density Lipoprotein (LDL) cholesterol, Total Cholesterol and Triglycerides will be assessed using clinical chemistry tests
Circulating Glucose | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  Glucose
Circulating Insulin | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  Insulin
Circulating Markers for Lysosomal Damage | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  Markers for lysosomal damage (cathepsin-D and acid-phosphatase)
Circulating Markers for Liver Health (1) | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  Alanine Aminotransferase (ALT) level will be determined using clinical chemistry
Circulating Markers for Liver Health (2) | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  Aspartate Transaminase (AST) level will be determined using clinical chemistry
Circulating Markers for Liver Health (3) | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  Gamma-Glutamyl Transferase (GGT) level will be determined using clinical chemistry
Circulating Markers for Liver Health (4) | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  Bilirubin level will be determined using clinical chemistry
Circulating Markers for Liver Health (5) | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  Cytokeratin-18 (CK-18) level will be determined using clinical chemistry
Single Nucleotide Polymorphisms (SNPs) | Change in outcomes at baseline before a 16-week skin roasted peanut intervention and 16-week control period.
  DNA from leucocytes will be analyzed for the presence of known SNPs in genes encoding proteins known to play a role in cholesterol metabolism.
Structural Brain Status | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  High-resolution anatomical MPRAGE scan
Fat Distribution in Abdomen | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  Magnetic Resonance Imaging measurements will be included to quantify abdominal fat compartments (i.e. subcutaneous and visceral fat)
Fat Content in Liver | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  Magnetic Resonance Imaging measurements will be included to quantify liver fat content
Other perceivable benefits: Quality of Life | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  The Quality of life will be assessed using a 32-item questionnaire
Other perceivable benefits: Sleep Characteristics | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  Sleep characteristics will be assessed using the 10-item Pittsburgh Sleep Quality Index
Other perceivable benefits: Mood | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  Mood will be tested using the Affect Grid
Other perceivable benefits: Stress | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  Stress will be assessed using the Perceived Stress Scale (PSS)
Other perceivable benefits: Physical Fitness (1) | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  Timed up-and-go test (TUGT)
Other perceivable benefits: Physical Fitness (2) | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  The 6-minute walk test (6 MWT)
Other perceivable benefits: Physical Fitness (3) | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  Handgrip test
Weight | Change in outcomes will be compared at baseline, at 8-weeks and at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  Weight in kilograms
Waist Circumference | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  Waist circumference in centimeters
Hip Circumference | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  Hip circumference in centimeters
Indirect Fat Distribution | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  Measured by skinfold measurements
Food Intake | Change in outcomes at the end of a 16-week skin roasted peanut intervention and 16-week control period.
  Food intake will be assessed using the Food Frequency Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Joris, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Kerkhof L, Mensink RP, Plat J, Nijssen KMR, Joris PJ. Longer-term skin-roasted peanut consumption improves brain vascular function and memory: A randomized, single-blind, controlled crossover trial in healthy older adults. Clin Nutr. 2025 Dec;55:170-179. doi: 10.1016/j.clnu.2025.10.020. Epub 2025 Nov 1. PMID 41205298